CLINICAL TRIAL: NCT01550575
Title: Patient Retrospective Outcomes (PRO)
Acronym: PRO
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A7005
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients eligible for SCS, RF or other treatment approaches: Patients who have previously been implanted with, or are eligible for implantation with a spinal cord stimulation system or various other treatment approaches such as RF, IDS, etc.
  Interventions: Device: Non Boston Scientific Systems; Device: Boston Scientific Systems
- Patients Eligible for treatment options with prior treatment: Patients who have previously been implanted with a spinal cord stimulation system or other various treatments, and have thereafter received a different form of chronic pain treatment such as a different SCS system, RF, IDS etc.
  Interventions: Device: Non Boston Scientific Systems; Device: Boston Scientific Systems

INTERVENTIONS:
Device: Non Boston Scientific Systems — Spinal cord stimulation, RF, IDS etc.
Device: Boston Scientific Systems — Spinal cord stimulation, RF, IDS etc

SUMMARY:
This study will evaluate de-identified (anonymous) data in subject medical charts to review the clinical outcomes of various treatment approaches in the treatment of chronic pain.

DETAILED DESCRIPTION:
This study is a retrospective, multi-center, de-identified patient data review.

The study will include multiple independent cohorts to evaluate clinical outcomes in different subgroups.

ELIGIBILITY:
Key Inclusion Criteria:

* Previously treated with or eligible for use with Boston Scientific Systems
* 18 years of age or older at the start of Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have previously been implanted with, or who are candidates for implantation with a spinal cord stimulation system or other various treatment approaches, such as radio frequency ablation or indirect decompression system (IDS).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2012-04-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Responder rate | Through study completion, approximately two years
  Responder rate for pain relief through study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (143):
- United States (87):
  - Lakeside Spine & Pain, Lake Havasu City, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Kern Neuroscience Institute, Bakersfield, California
  - Pain Consultants of San Diego, Chula Vista, California
  - Pain Medicine Associates, Inc., Fountain Valley, California
  - UCSD Medical Center - Jacobs Medical Center, La Jolla, California
  - California Orthopedics & Spine, Larkspur, California
  - MarinHealth Spine Institute, Larkspur, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Newport Beach Headache and Pain, Newport Beach, California
  - Vitamed Research, Rancho Mirage, California
  - Pacific Pain Management, Inc., Ventura, California
  - IPM Medical Group Inc., Walnut Creek, California
  - Barolat Neuroscience, Denver, Colorado
  - Advanced Diagnostic Pain Treatment Centers, New Haven, Connecticut
  - Orlando Health Neuroscience Institute, Clermont, Florida
  - Florida Spine Specialists, Fort Lauderdale, Florida
  - Louis J. Raso, MD, PA, Jupiter, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - Advanced Interventional Pain Management and Research Clinic, Inc., Miami Gardens, Florida
  - Florida Pain Clinic, Ocala, Florida
  - Orthomicrospine, Pensacola, Florida
  - HCA Florida West Orthopedic Specialists, Pensacola, Florida
  - West Florida Orthopedics and Spine Surgery, Pensacola, Florida
  - Interventional Spine and Pain Institute, Vero Beach, Florida
  - Orthopedic Research Foundation, Savannah, Georgia
  - Centurion Spine and Pain, Waycross, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Pain and Spine Specialists of Idaho, Idaho Falls, Idaho
  - North Idaho Day Surgery, Post Falls, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Summit Research Institute, Fort Wayne, Indiana
  - Comprehensive Pain and Spine Specialists, Muncie, Indiana
  - Henry Community Health, New Castle, Indiana
  - Precision Spine Care, Overland Park, Kansas
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Pain and Spine Specialist of Maryland, Mount Airy, Maryland
  - Michigan Orthopedic Center, Lansing, Michigan
  - Multidisciplinary Pain Management Services, Okemos, Michigan
  - Forest Health Medical Center, Ypsilanti, Michigan
  - Twin Cities Pain Clinic & Surgery Center, Edina, Minnesota
  - NeuroSpecs-Gulfport Performance Spine, Gulfport, Mississippi
  - Comprehensive Pain & Rehabilitation, Pascagoula, Mississippi
  - Saint Louis Pain Consultants, Chesterfield, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Albany Medical Center, Albany, New York
  - Jeffrey M. Epstein, M.D. PC, Babylon, New York
  - Montefiore Medical Center, The Bronx, New York
  - Spine and Skeletal Pain Medicine, Utica, New York
  - Integrative Pain and Wellness Associates, Williamsville, New York
  - Vidant Roanoke - Chowan Hospital Pain Center, Ahoskie, North Carolina
  - Carolinas Research Institute, PLLC, Huntersville, North Carolina
  - Crystal Coast Pain Management, New Bern, North Carolina
  - Piedmont Interventional Pain Care, Salisbury, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Interventional Pain and Spine, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Orthopaedic and Spine Center, Dublin, Ohio
  - Cincinnati Comprehensive Pain Center, Fairfield, Ohio
  - Western Reserve Spine and Pain Institute, Kent, Ohio
  - Interventional Pain Consultants, Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Pain Specialists of Southern Oregon, Medford, Oregon
  - Quave Clinic, Medford, Oregon
  - Southern Oregon Orthopedics, Medford, Oregon
  - Summit Spine, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Florence Neurosurgery and Spine, Florence, South Carolina
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Interventional Spine and Pain Center, Manchester, Tennessee
  - Comprehensive Pain & Neurology Center, Murfreesboro, Tennessee
  - Pain Center Physicians, Austin, Texas
  - Balcones Pain Consultants, Austin, Texas
  - KSF Orthopaedics, Houston, Texas
  - Central Texas Pain Institute, Killeen, Texas
  - Advanced Spine Pain Solutions, Laredo, Texas
  - Spine Team Texas, Southlake, Texas
  - Space City Pain Specialists, Webster, Texas
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - EvergreenHealth Pain Care, Kirkland, Washington
  - Mind Your Body Institute, Seattle, Washington
  - Northwest Pain Care, Spokane, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Interventional Pain Specialists of Wisconsin, Rice Lake, Wisconsin
- Australia (8):
  - Berwick Pain Management, Berwick
  - Hunter Pain Clinic, Broadmeadow
  - Monash Clinical Research, Caulfield South
  - Green Lizard Science, Claremont
  - Sydney Spine and Pain Pty Ltd, Hurstville
  - Sunshine Coast Clinical Research, Noosa
  - Womens Health and Research Institute of Australia, Sydney
  - Pain Medicine of South Australia, Wayville
- Clinique Saint-Pierre Ottignies, Ottignies, Belgium
- France (7):
  - Polyclinique du Parc, Caen
  - Clinique de la Sauvegarde, Lyon
  - Hopital Prive du Confluent SAS, Nantes
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHU La Miletrie, Poitiers
  - CHU de Nantes-Hopital Laennec, Saint-Herblain
  - Hopital Foch, Suresnes
- Germany (5):
  - Inter Neuro, Berlin
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - St. Marien-Hospital Hamm, Hamm
  - University Berlin, Charite Virchow Standort, Wedding, Wedding
- Italy (7):
  - Pres. Osp. Civile Santi Antonio e Biagio, Alessandria
  - Az. Osp. Monaldi, Napoli
  - AUSL della Romagna, Ravenna
  - Ospedale San Giuliano, Rionero in Vulture
  - Ospedale S. Giovanni Addolorata, Rome
  - Policlinico Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Netherlands (2):
  - Alrijne Ziekenhuis Leiderdorp, Leiderdorp
  - Ziekenhuis Rijnstate, Velp
- CHU Sao Joao, Porto, Portugal
- Ponce Interventional Pain Center, Ponce, Puerto Rico
- Spain (15):
  - Hospital De Bellvitge, Barcelona
  - H. Puerta Del Mar, Cadiz
  - Complejo Hospitalario Universitario de Cartagena, Cartagena
  - Hospital Universitario Doctor Jose Molina Orosa, Las Palmas
  - Hospital San Pedro, Logroño
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Quiron Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Complexo Hospitalario Universitario de Ourense (CHUO), Ourense
  - Hospital Virgen Del Rocio, Seville
  - H. Clinico Universitario, Valencia
  - Hospital de la Ribera, Valencia
  - Hospital Universitario La Fe, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Switzerland (2):
  - La Tour Hospital, Meyrin
  - Ospedale Regionale di Lugano, Viganello
- United Kingdom (6):
  - Basildon and Thurrock University Hospitals NHS, Basildon
  - Southmead Hospital Bristol, Bristol
  - Royal Devon & Exeter Hospital, Exeter
  - The General Infirmary, Leeds
  - St. Bartholomews Hospital, London
  - James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Ferro R, North J, Kranenburg A, Pyles S, Dorenkamp C, Poston J, Schneider J, Auten K, Goldberg E. Automated Neural Dosing for Fast-Acting Subperception Therapy: Sustained Spinal Cord Stimulation Outcomes from a Multicenter Study. Pain Ther. 2025 Aug;14(4):1417-1429. doi: 10.1007/s40122-025-00758-y. Epub 2025 Jul 3. PMID 40603812
- [Derived] Metzger C, Hammond B, Ferro R, North J, Pyles S, Kranenburg A, Washabaugh E, Goldberg E. Two-year outcomes using fast-acting sub-perception therapy for spinal cord stimulation: results of a real-world multicenter study in the United States. Expert Rev Med Devices. 2025 Jan-Feb;22(2):155-164. doi: 10.1080/17434440.2025.2453554. Epub 2025 Jan 16. PMID 39819320